CLINICAL TRIAL: NCT02584972
Title: Postural Control During Walking and Standing Among Children With Autism Spectrum Disorder
Acronym: PCASD
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Itshak Melzer, Associate professor, Soroka University Medical Center
Other Study IDs: Sor 274-13 CTIL
Record Dates: First submitted 2015-10-18; First posted 2015-10-23 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Postural control; Gait; Children; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- children with Autism Spectrum Disorder: no intervention required
  Interventions: Other: no intervention required
- heathy children: no intervention required
  Interventions: Other: no intervention required

INTERVENTIONS:
Other: no intervention required — no intervention required

SUMMARY:
Lately, many researchers have found that Children with autism spectrum disorder (ASD) are most likely to have gross motor deficiencies such as lack of coordination in gait and balance. Much has been researched on etiology and motor learning, but only very few researches have examined and analyzed quantitatively gait and balance in ASD. The aim of this research is to analyze quantitatively balance, gait and balance during perturbation in children with ASD and to compare with typically developed children (TD). A group of 20 children diagnosed with ASD and a control group of 20 TD children will be recruited and tested in the laboratory with well-established measures of gait and balance function. They will be instructed to stand as still as possible on a force plate with different task conditions : (1) standing with the eyes open (EO) - standing upright viewing an "X" displayed on a screen 3 meters in front of them; (2) eyes closed (EC) - same as (1) with the eyes closed and covered by blindfolds (i.e. no visual information). (3) Same as 1 standing on foam (i.e., conflicting proprioceptive information). Gait will be measured using the narrow base walk test, modified for clinical use. Participants will be asked to walk within a narrow path 6 meters long . The statistical analysis will include Independent T-tests to compare the ASD and controls with respect to different characteristics. General Linear Model (GLM) will be used by applying a separate model where the dependent variables will be the average values of the postural stability or gait stability parameters (continuous) and the independent variables were categorical by the group and task condition.

DETAILED DESCRIPTION:
Study protocol The study group will be consisted of 30 ASD children (6-12 years old) who were diagnosed with ASD recruited in the Pediatric Neurology clinic at Soroka Medical Center, Beer-Sheva, Israel, and ASD centers. A convenience sample of 30 age-gender matched healthy control children (6-12 years old) will be recruited using ads and flayer in Beer-Sheva and area. Children's parents will sign the informed consent, in accordance with procedures approved by the Helsinki Ethics Committee in Soroka Medical Center. As part of the initial assessment all children including the control group subjects will undergo a complete neuro-developmental and motor screening evaluation by an experienced pediatric neurologist using the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnostic criteria Children with autism have to meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria. ASD participants will have to communicate enough in order to cooperate and understand orders. Exclusion criteria are: ASD children who were diagnosed with neurological, orthopedic, or psychiatric diagnoses according to DSM-IV criteria that can affect motor control and postural stability; cerebral palsy; neuropathic diseases; limb fracture; head trauma during the previous year; use of any medication other than MPH during the study period; and who had an IQ score below the normal range (<70), as assessed by the Wechsler Intelligence Scale for Children - Revised (Wisc-R) administered by a child psychologist.

Recruitment procedure ASD participants will be recruited in the children neurology department at Soroka Medical center. Control group subjects will be recruited from the community using personal contacts using ads and flayer. The PI of this project (Prof. Zamir) will not be involved in the recruitment procedure of the children's under his clinical practice.

Outcome Assessments: Postural stability Protocol The assessment procedure will be made in the ediatric Neurology clinic at Soroka Medical Center, Beer-Sheva, the parents will sign of the informed consent than the participant will be instructed to stand upright as still as possible on the force platform with the feet positioned as close as possible (heels and toes touching). A total of five 30-second quiet-standing trials will be obtained from each participant instructed to stand as still as they possibly can in two task conditions. Two minute rest break will be provided between two task conditions and thirty seconds rest breaks between the trials. The two task conditions are: (1) standing with the eyes open (EO) - standing upright viewing an "X" displayed on a screen 3 meters in front of them; (2) eyes closed (EC) - same as (1) with the eyes closed and covered by blindfolds (i.e. no visual information). (3) Same as 1 standing on foam (i.e., conflicting proprioceptive information). Balance measurements will be collected with a Kistler 9287 single force platform (Kistler Instrument Corp., Winterthur, Switzerland) that measures the time-varying displacement of the Center of pressure (CoP). The force platform data will be sampled at a frequency of 100 Hz and stored on a hard disk for later processing. Four well-established parameters of postural stability will be extracted using automatic code written in Matlab (Math Works Inc., Cambridge, MA, USA): 1) Mediolateral CoP range (mm) (ML-sway Range); 2) Anterioposterior CoP range (mm) (AP-sway Range); 3) Mean velocity of CoP sway (mm/sec); 4) Sway area (mm2) - the elliptical area of the CoP points. Lower postural stability scores indicate higher levels of postural control. Also four parameters of SDA were extracted using automatic code written in Matlab: 1) short-term diffusion coefficients in mm2s-1 (Drs); 2) long-term diffusion coefficients in mm2s-1 (Drl); 3) the Critical Time in sec (Ctr); and 4) Critical Displacement in cm (Cdr). These parameters will be computed for each subject's trials, and then averaged for each set of 5 trials to obtain an average value for each parameter and for each subject, in each experimental condition.

Gait stability protocol After a 10-minute break, gait will be measured using the narrow base walk test, modified for clinical use. Participants will be asked to walk within a narrow path (6 meters long) first without and then with a concurrent cognitive task (ST- and DT), always in the same order. The test incorporates measurement of lateral instability during gait. The width of the narrow path will be normalized to 50% of the distance between the participant's anterior superior iliac spines + the width of the subject's shoe. This produces a similar challenge for individuals with different body morphologies. The narrow path will be outlined by two narrow six meter black mattresses on the walking surface; the participants will be instructed to walk within the path without stepping on the black mattresses. All trials will be videotaped using a video-camera that was placed 2 meters in front of the walking path and 1.5 meters high to detect trial time and step errors during the test. Step error is defined as every step where the subject's shoes step outside the narrow path, touching the black mattresses outlining the sides of the narrow base walkway. test-re-test agreement of NBWT found to be high for all variables; ICC(1,2) 0.77-0.92 in ST and 0.78-0.92 in DT (unpublished data).

ELIGIBILITY:
Inclusion Criteria:

* children with autism spectrum disorder
* 6-12 years old
* able to walk independently

Exclusion Criteria:

* ASD children who were diagnosed with neurological, orthopedic, or psychiatric diagnoses according to DSM-IV criteria that can affect motor control and postural stability;
* cerebral palsy; - neuropathic diseases;
* limb fracture;
* head trauma during the previous year;
* who had an IQ score below the normal range (<70), as assessed by the Wechsler Intelligence Scale for Children - Revised (Wisc-R) administered by a child psychologist.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with autism spectrum disorder
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
postural stability measures | baseline

SECONDARY OUTCOMES:
6 meter Narrow Path Walking Test | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Itshak Melzer, Phd, Principal Investigator — Ben-Gurion University of the Negev
Locations (2):
- Israel (2):
  - Ben-guion University of the Negev,, Beersheba
  - Soroka University Medical Center, Beersheba